CLINICAL TRIAL: NCT00218166
Title: GABA Agonists as Pharmacotherapies for Cocaine Abuse
Brief Title: Effectiveness of GABA Agonists in Reducing the Reinforcing Effects of Cocaine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Craig R. Rush, University of Kentucky
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: DA013567; R01-13567-1; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-10

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine; tiagabine; baclofen
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — GABA Agonists; Triazolam; Tiagabine; Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (No Intervention): Within subject design
  Interventions: Drug: GABA Agonists

INTERVENTIONS:
Drug: GABA Agonists — GABA drugs administered acutely by mouth
  Other Names: Triazolam, tiagabine, baclofen

SUMMARY:
Cocaine abuse continues to represent a significant public-health concern. Cocaine likely creates its addictive effects by increasing levels of dopamine, a chemical found in the brain. GABA agonists are chemicals that have the opposite effect of cocaine by inhibiting the release of dopamine. The purpose of this study is to determine whether GABA agonists reduce the psychological and physiological reinforcing effects of cocaine.

DETAILED DESCRIPTION:
Cocaine likely creates its reinforcing and addictive effects by increasing levels of dopamine, a brain neurotransmitter. GABA agonists are chemicals that have the opposite effect by inhibiting the release of dopamine. Increasing GABA activity may result in greater inhibition of dopamine systems, which may lead to new treatments for cocaine abuse. The purpose of this study is to determine whether pretreatment with GABA agonists reduces the psychological and physiological reinforcing effects of cocaine. Specifically, the study will look at three different GABA agonists: tiagabine, baclofen, and trazolam.

This double-blind, placebo-controlled study will involve three separate experimental phases; each phase will last 4 weeks and will test one of three GABA agonists (tiagabine, baclofen, or trazolam). Daily testing sessions will last approximately 6 hours. One of four GABA agonist dose treatments will be administered. Participants will then be introduced to a sample dose of intranasal cocaine. This will allow the participants to become acquainted with the drug effects of the corresponding cocaine dose for that day (0.444, 5, 10, or 20 mg). Subjective, physiological, and performance measures will be obtained. This will be followed by a period of cocaine self-administration. Participants will be given the opportunity to work on a computer to obtain additional single unit doses of cocaine. A total of 8 unit doses of cocaine will be available during each daily session. At the end of the daily session, additional subjective measures will be evaluated with questionnaires. Overall, a total of 16 GABA agonist-cocaine dose combinations will be administered on 16 different days. A subgroup of participants will also undergo similar procedures with the option to acquire money instead of cocaine. At the end of the study, all participants will be offered a referral to an appropriate drug-abuse treatment program.

ELIGIBILITY:
Inclusion Criteria:

* Recent use of cocaine
* Meets DSM-IV diagnostic criteria for psychoactive substance abuse or dependence for cocaine
* Positive drug urine screen for cocaine at time of initial screening interview
* Reports self-administration of at least 1,260 mg of cocaine during the 4 weeks prior to study start date
* Body Mass Index (BMI) of less than 29
* Females must use an effective form of contraception throughout the study

Exclusion Criteria:

* Meets DSM-IV diagnostic criteria for psychoactive substance dependence for substances other than cocaine or nicotine
* Currently seeking treatment for substance abuse/dependence
* Current or past history of physical disease, impaired cardiovascular functioning, chronic obstructive pulmonary disease
* History of seizure, head traumas, or central nervous system tumors
* Current or past history of serious psychiatric disorder other than substance abuse or dependence
* Family history of cardiovascular disease or seizure disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2001-08; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Progressive-ratio break point | Measured during each experimental session

SECONDARY OUTCOMES:
Subjective effects of cocaine | Measured during each experimental session
Physiological measures | Measured throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Craig Rush, Principal Investigator — ACT
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States